CLINICAL TRIAL: NCT06601777
Title: Evaluation of the Effectiveness, Safety, and Cost of a Smart Hospital System for Patients With Chronic Obstructive Pulmonary Disease: Prospective Multicenter Randomized Controlled Trial
Brief Title: Evaluation of the Effectiveness, Safety, and Cost of a Smart Hospital System for Patients With Chronic Obstructive Pulmonary Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 4-2024-0299
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The Smart Homespital system can be applied for the first 3 months (12 weeks), and then the primary and secondary variables will be evaluated at 3, 6, 9months.
  Interventions: Behavioral: Immediate application of the Smart Homespital system
- attention-waitlist control group (Experimental): The waiting list-control group will receive general medical services for the first 3 months and will receive the Smart Homespital system for 3-6 months. Primary and secondary variables will be evaluated between 3, 6, and 9 months.
  Interventions: Behavioral: Delayed application of the Smart Homespital system after 3 months

INTERVENTIONS:
Behavioral: Immediate application of the Smart Homespital system — The Smart Homespital system can be applied for the first 3 months (12 weeks), and then the primary and secondary variables will be evaluated at 3, 6, 9months. While applying the Smart Homespital system, exercise three times a week, measure sleep twice a week, and questionnaire assessments (mMRC, CRQ, EQ-5D, K-CESD) are conducted once every two weeks.
  Arms: intervention group
Behavioral: Delayed application of the Smart Homespital system after 3 months — The waiting list-control group will receive general medical services for the first 3 months and will receive a Smart Homespital system for 3-6 months. Primary and secondary variables will be monitored between 3, 6, and 9 months. While applying the Smart Homespital system, exercise three times a week, measure sleep twice a week, and questionnaire assessments (mMRC, CRQ, EQ-5D, K-CESD) are conducted once every two weeks.
  Arms: attention-waitlist control group

SUMMARY:
This study aims to analyze the effectiveness/safety/cost of the Smart Homespital system that provides a service that allows patients with Chronic Obstructive Pulmonary Disease to easily access and use biosignals generated using biosignal collection medical equipment at home.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with COPD who meet the following pulmonary function test results:

1. Pre FEV1 < 80% **or**
2. Pre FVC < 80% **or**
3. DLCO < 60%

Exclusion Criteria:

1. Patients who do not agree to participate in the study.
2. Patients who fail to use the medical device equipment.
3. Patients where tracking during the study period is expected to be impossible.
4. Patients who have difficulty communicating verbally.
5. Patients who are bedridden or unable to exercise at all due to severe cardiorespiratory dysfunction.
6. Patients receiving hospital-centered rehabilitation treatment during the study period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Respiratory symptom questionnaire | After applying the Smart Homespital system(12weaks)
  For survey scores, success is defined as an increase in the respective defined MCID(the minimal clinically important difference) rises the baseline.
  1) Chronic respiratory questionnaire (CRQ)
  * Success: 4 points or more 2.)Modified Medical Research Council dyspnea scale (mMRC)
  * Success: 1points or more 3) EQ-5D
  * Success: 1 points or more

SECONDARY OUTCOMES:
Depression Questionnaire | Survey every 2 weeks during the 12-week Homespital system application, then at 3, 6, and 9 months after the start of the study.
  K-CESD-R : Survey every 2 weeks during the 12-week Homespital system application, then at 3, 6, and 9 months after the start of the study.
  * Success Criteria: Achieving 4 points or more.
  * Success: 4 points or more
Service satisfaction evaluation | After 12 weeks of applying the Smart Homespital system.
  CSQ-8: After 12 weeks of applying the Smart Homespital system.
  - Success Criteria: Achieving 4 points or more.
safety | Measured after the study ends (9 months later).
  * Number of hospital visits directly related to the Smart Home Hospital Program
  * Success Criteria: Less than 2 hospital visits related to the Smart Homespital program.
cost assessment | After study ends (9 months later)
  Criteria: Comparison of average hospital respiratory rehabilitation treatment costs with the Smart Homespital program's costs.
6 minute walking test | At 3, 6, and 9 months.
  - Success Criteria: More than a 10% increase over the baseline.
pulmonary function test | At 3, 6, and 9 months.
  Success Criteria: Increase in FVC, FEV1, or DLCO by more than 10% at the time of registration.
system compliance | During the 12-week period of applying the Homespital system.
  Criteria: Maintaining a minimum of 5,000 steps/day during the 12-week period of applying the Homespital system.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No